CLINICAL TRIAL: NCT06611332
Title: Efficacy and Safety of Electroacupuncture on Lumbar Disc Herniation with Radiculopathy: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Electroacupuncture on Lumbar Disc Herniation with Radiculopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhou, Professor, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: JXUCM-ACU-01
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Lumbar Disc Herniation; Radiculopathy Lumbar
Keywords: electroacupuncture; radiculopathy; sham control; randomized controlled trial; lumbar disc herniation
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electroacupuncture (Experimental)
  Interventions: Other: Electroacupuncture
- Sham electroacupuncture (Sham Comparator)
  Interventions: Other: Sham electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — The main acupoints selected for the electroacupuncture group are bilateral BL23, bilateral BL25, bilateral GB30, bilateral LR11, bilateral LR8, GV4, GV3, and the affected BL40, and the secondary acupoints selected are bilateral BL54, the affected side BL57 and the affected side BL60.The treatment will be administered once every other day for 30 minutes each time, lasting for 8 consecutive weeks, totaling 24 sessions.
  Arms: Electroacupuncture
Other: Sham electroacupuncture — In the sham electroacupuncture group, the acupoints will be at a position 2 cm lateral to the correct acupoints horizontally. The dosage and treatment course are the same as those in the electroacupuncture group.
  Arms: Sham electroacupuncture

SUMMARY:
Lumbar disc herniation with radiculopathy (LDHR) is the local displacement of the intervertebral disc and its contents beyond the edge of the normal intervertebral disc space, resulting in pain, weakness or numbness in the muscle or dermatomal distribution area. Electroacupuncture is based on obtaining the needling sensation manually and applying electrical stimulation of different frequencies and intensities, aiming to enhance the intensity of acupoint stimulation to improve the effect. As a kind of acupoint stimulation therapy, electroacupuncture has shown analgesic effects in animal experiments. However, at present, the clinical evidence of electroacupuncture applied in the treatment of LDHR is still insufficient. Therefore, this randomized, single-blind, sham electroacupuncture controlled trial aims to evaluate the efficacy and safety of electroacupuncture as a treatment for LDHR.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 70 years old.
2. With intervertebral disc protrusion confirmed by a MRI or CT, accompanied by radicular pain in the lower extremities.
3. With a NRS score ≥ 4 points for both low back pain and leg pain, and the pain lasts for at least 3 months;
4. Voluntarily participating the trial and signing the informed consent form.

Exclusion Criteria:

1. Previous surgical treatment of the spine.
2. Received any physical therapy for lumbar disc herniation within the recent 3 months.
3. Complicated with diseases that can cause low back and leg pain.
4. Symptomatic foraminal stenosis caused by severe degenerative diseases, accompanied by severe nerve injuries.
5. Previous severe mental illness, organ failure, or malignant tumor.
6. Planned spinal surgery or other major surgeries within the next 3 months.
7. Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders | Weeks 8 and 24
  Definition of a response: a reduction of at least 2 points in the score of the Numerical Rating Scale for both low back pain and leg pain.

SECONDARY OUTCOMES:
Intensity of low back pain | Weeks 2, 4, 8, 16, and 24
  Changes from baseline in the intensity of low back pain assessed by the Numerical Rating Scale
Intensity of leg pain | Weeks 2, 4, 8, 16, and 24
  Changes from baseline in intensity of leg pain assessed by the Numerical Rating Scale
Level of disability | Weeks 2, 4, 8, 16, and 24
  Changes from baseline in the level of disability assessed by the Roland-Morris Disability Questionnaire
Performance status | Weeks 2, 4, 8, 16, and 24
  Changes from baseline in functional status assessed by the Japanese Orthopaedic Association Score
Severity of depression | Weeks 2, 4, 8, 16, and 24
  Changes from baseline in the severity of depression assessed by the Hamilton Depression Rating Scale
Severity of anxiety | Weeks 2, 4, 8, 16, and 24
  Changes from baseline in the severity of anxiety assessed by the Hamilton Anxiety Rating Scale
Sleep quality | Weeks 2, 4, 8, 16, and 24
  Changes from baseline in sleep quality assessed by the Insomnia Severity Index
Pain self-efficacy | Weeks 2, 4, 8, 16, and 24
  Changes from baseline in pain self-efficacy assessed by the Pain self-efficacy questionnaire
Use of analgesics | Weeks 8 and 24
  The proportion of patients who used analgesics for emergency.
Incidence of lumbar spine surgery | Weeks 8 and 24
  The incidence of lumbar spine surgery during the follow-up
Incidence of any adverse events | Weeks 8 and 24
  Adverse events be reported by patients and determined by clinicians.
Incidence of treatment-related adverse events | Weeks 8 and 24
  Treatment-related adverse events include adverse events caused by electroacupuncture or sham electroacupuncture treatment.
Incidence of serious adverse event | Weeks 8 and 24
  Serious adverse events refer to adverse events that require hospitalization or an extended hospital stay, result in disability, pose a threat to life, or cause death.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Jiangxi University of Chinese Medicine, Jiangxi, Nanchang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Liu L, Yuan L, Liu X, Ding H, Zhou X, Cao Q. A Randomized, Sham-Controlled Trial on the Efficacy and Safety of Electroacupuncture for Lumbar Disc Herniation with Radiculopathy: Rationale and Study Protocol. J Pain Res. 2025 May 5;18:2307-2319. doi: 10.2147/JPR.S512711. eCollection 2025. PMID 40352817